CLINICAL TRIAL: NCT01144962
Title: Allogeneic Bone Marrow Derived Mesenchymal Stem Cells for the Treatment of Fistulas in Patients With Refractory Perianal Crohn's Disease
Brief Title: Dose-escalating Therapeutic Study of Allogeneic Bone Marrow Derived Mesenchymal Stem Cells for the Treatment of Fistulas in Patients With Refractory Perianal Crohn's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: DigestScience (Unknown)
Responsible Party: Principal Investigator, HeinVerspaget, Professor, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P10.102
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Crohn's Disease; Fistula
Keywords: Crohn's Disease; Fistula; Mesenchymal Stem Cell; Mesenchymal Stromal Cell; MSC; IBD
MeSH Terms: conditions — Crohn Disease; Fistula

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control group (Sham Comparator): Patients in the control group will undergo surgical localization, curettage of the fistulous tract and closure of the internal opening, without injection of MSCs.
  Interventions: Procedure: Localization, curettage of the fistulous tract and closure of the internal opening without MSC injection.
- Cohort 1 (Active Comparator): 10x10^6 MSC
  Interventions: Procedure: Localization, curettage of the fistulous tract and closure of the internal opening with local MSC injection.
- Cohort 2 (Active Comparator): 30x10^6 MSC
  Interventions: Procedure: Localization, curettage of the fistulous tract and closure of the internal opening with local MSC injection.
- Cohort 3 (Active Comparator): 90x10^6 MSC
  Interventions: Procedure: Localization, curettage of the fistulous tract and closure of the internal opening with local MSC injection.

INTERVENTIONS:
Procedure: Localization, curettage of the fistulous tract and closure of the internal opening without MSC injection. — Patients will undergo surgical localization, curettage of the fistulous tract and closure of the internal opening, without injection of MSCs.
  Arms: Control group
Procedure: Localization, curettage of the fistulous tract and closure of the internal opening with local MSC injection. — Patients will undergo surgical localization, curettage of the fistulous tract and closure of the internal opening, with local injection of indicated dose of MSCs
  Arms: Cohort 1; Cohort 2; Cohort 3

SUMMARY:
In a dose escalation study we will determine the safety and preliminary efficacy of allogeneic bone marrow mesenchymal stem cells (bmMSCs) in the induction of response for active fistulizing Crohn's Disease (CD).

DETAILED DESCRIPTION:
Despite the introduction of anti-TNFa (tumor necrosis factor alpha) therapy, perianal disease still accounts for a high rate of morbidity in patients diagnosed with CD. Recently, a phase II multicenter randomized study was reported showing that expanded adipose tissue derived mesenchymal stem cells (atMSCs) in combination with fibrin glue was an effective and safe treatment for complex perianal fistula. However, dose escalation of allogeneic bone marrow (bm) MSCs for the local treatment of perianal fistulas has not been studied.

In this study, three escalating doses will be tested in a total of three cohorts. MSC implantation will be preceded by surgical localization, curettage of the fistulous tract and closure of the internal opening. Per cohort, patients will be randomized in a 5:2 fashion to receive either 10x10^6 (cohort 1), 30x10^6 (cohort 2) or 90x10^6 (cohort 3) bmMSCs or no cells (control group).

The primary endpoint will be assessed at week 12: i) the number of adverse and serious adverse events and ii) a reduction in the number of draining fistulas, which is defined as absence of discharge and absence of collections of ≥2 cm directly related to the treated fistulas tracts as measured by MRI.

ELIGIBILITY:
Inclusion Criteria:

* Men and women > 18 years of age
* Patient must have had CD (for at least 3 months from the time of initial diagnosis). The diagnosis of CD must have been confirmed by endoscopic and histologic evidence
* CDAI score of <250 at screening and baseline
* Peri-anal fistulas must be refractory to conventional medical therapy Which means that at some time during the course of the disease, patient must have received both steroids and immunosuppressive agents (for example, azathioprine, 6-mercaptopurine (6-MP), methotrexate, or infliximab) which did not result in an adequate response to treatment
* Patients with previous surgical attempts to eradicate perianal fistulas are eligible for inclusion as are patients with setons in situ. Setons will be removed during the surgical procedure
* Patients included in the study might be receiving 5-aminosalicylic acid (5-ASA), steroids, azathioprine, 6-MP, methotrexate, or any similar drug at the time of enrolment and is allowed to have a history of infliximab treatment, provided the following conditions are fulfilled at screening:
* The dose of 5-ASA (both oral and rectal) must have been stable for at least 4 weeks prior to enrollment
* The dose of steroids must be stable for at least 4 weeks prior to enrollment
* The dose of immunosuppressants (for example azathioprine, 6-MP, or methotrexate) must have been stable for at least 8 weeks prior to enrollment and the patient on therapy for at least three months prior to enrollment
* The last dose of infliximab or other anti-TNF drug is > 8 weeks prior to enrollment
* No need for immediate surgery (obstruction, strictures or abscess)
* If female and of child-bearing age, patient must be non-pregnant non-breastfeeding, and use adequate contraception
* Patient is willing to participate in the study and has signed the informed consent. Consent must be obtained prior to any study procedure

Exclusion Criteria:

* Patients with evidence of acute peri-anal infection, presence of peri-anal abscesses larger than 2 cm, and anal or rectal stricture
* Patients with evidence of any infections needing antibiotic treatment
* Rectovaginal fistulas, or complex peri-anal fistulas with more than two internal openings
* Patients suffering from renal- or hepatic failure
* Use of any investigational drug within 1 month prior to screening or within 5 half-lives of the investigational agent, whichever is longer
* Patient is allergic to gadolinium (MRI contrast agent)
* Patient with severe renal insufficiency defined as patients with a glomerular filtration rate (GFR) below 60 mL/min/1.73 m2. GFR = 186.3 x (serum creatinine)-1.154 x (age in years)-0.203 x 1.212 (if patient is black) x 0.742 (if female)
* Due to the high strength electromagnetic fields that will be used during MRI there is a risk of interference with any metallic implants in the body. The following conditions will disqualify patients from having an MRI and will be excluded from this study:

  * Electronically, magnetically, and mechanically activated implants
  * Ferromagnetic or electronically operated stapedial implants
  * Cardiac pacemakers/carotid sinus pacemaker implant
  * Hemostatic clips
  * Metallic splinters in the orbit
  * Insulin pumps and nerve stimulators
  * Lead wires or similar wires
  * Metal intrauterine device
* Change in concomitant medication:

  * Steroids must be stable for at least 4 weeks prior to enrollment
  * 5-ASA should be on a stable dose > 4 weeks prior to enrollment
  * Immunosuppressants (e.g. azathioprine, 6MP or methotrexate) should be on a stable dose > 8 weeks prior to enrolment
  * Infliximab or other anti-TNF antibody therapy should not be administered < 8 weeks prior to enrollment
* Claustrophobia
* Documented HIV (Human Immunodeficiency Virus) infection. Active hepatitis B, hepatitis C or TB
* Patients who currently have or who have had an opportunistic infection (e.g., herpes zoster [shingles], cytomegalovirus, Pneumocystis carinii, aspergillosis, histoplasmosis, or mycobacteria other than TB) within 6 months prior to screening
* Serious infections (such as pneumonia or pyelonephritis) in the previous 3 months. Less serious infections (such as acute upper respiratory tract infection [colds] or simple urinary tract infection) need not be considered exclusions at the discretion of the investigator
* Malignancy within the past 5 years (except for squamous or basal cell carcinoma of the skin that has been treated with no evidence of recurrence)
* History of lymphoproliferative disease including lymphoma
* Patient is unwilling or unable to comply with the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-06; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy (fistula closure) | 12 weeks
  i) the number of adverse and serious adverse events and ii) a reduction in the number of draining fistulas, which is defined as absence of discharge and absence of collections of ≥2 cm directly related to the treated fistulas tracts as measured by MRI (Magnetic Resonance Imaging).

SECONDARY OUTCOMES:
Clinical scores | 12 weeks
  1. To assess changes in the Crohn's Disease Activity Index (CDAI), the Perianal Disease Activity Index (PDAI) and the adapted Vaizey fecal incontinence score before and after mesenchymal stem cell (MSC) treatment;
Endoscopic scores | 12 weeks
  2. To compare endoscopic changes before and after local bmMSC treatment using the Crohn's Disease Endoscopic Index of Severity (CDEIS) and simplified endoscopic activity score for Crohn's disease (SES-CD);
Quality of life | 12 weeks
  3. To evaluate the effect of local treatment with autologous bmMSCs on the quality of life of patients with fistulizing CD using the short Inflammatory Bowel Disease Questionnaire (sIBDQ) and Short Form (SF)-36 score;
C-reactive protein (CRP) | 12 weeks
  4. To summarize the changes from baseline compared to 12 weeks in serum C-reactive protein (CRP).
Safety | 12 and 24 weeks
  5. To assess the incidence of surgical intervention and infections.

CONTACTS AND LOCATIONS:
Overall Officials: Hein W Verspaget, PhD, Study Chair — Leiden University Medical Center (LUMC)
Locations (1):
- Leiden University Medical Center (LUMC), Leiden, South Holland, Netherlands

REFERENCES:
- [Derived] Molendijk I, Bonsing BA, Roelofs H, Peeters KC, Wasser MN, Dijkstra G, van der Woude CJ, Duijvestein M, Veenendaal RA, Zwaginga JJ, Verspaget HW, Fibbe WE, van der Meulen-de Jong AE, Hommes DW. Allogeneic Bone Marrow-Derived Mesenchymal Stromal Cells Promote Healing of Refractory Perianal Fistulas in Patients With Crohn's Disease. Gastroenterology. 2015 Oct;149(4):918-27.e6. doi: 10.1053/j.gastro.2015.06.014. Epub 2015 Jun 25. PMID 26116801